CLINICAL TRIAL: NCT07343674
Title: PERFECT - Portuguese Evolut Registry Studying the Outcomes of Medtronic Evolut™ FX+ TAVI System by Evaluating an Optimal Care Pathway for TAVI
Acronym: PERFECT
Status: Not yet recruiting | Type: Observational
Sponsor: Portuguese Association of Interventional Cardiology (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PERFECT Registry
Record Dates: First submitted 2025-11-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Severe Symptomatic Aortic Stenosis (Defined as New York Heart Association (NYHA) Class ≥ II)
Keywords: TAVI; Transcatheter Aortic Valve Implantation; Evolut FX+; Aortic Stenosis; Cusp Overlap Technique; Conduction Disorders; Evolut FX+ TAVI System; TAVI System
MeSH Terms: conditions — Aortic Valve Stenosis; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients with severe aortic stenosis undergoing Medtronic Evolut FX+ TAVI System: Subjects with severe, symptomatic aortic stenosis (AS) with indication for TAVI (Transcatheter Aortic Valve Implant) with the Medtronic Evolut™ FX+ TAVI System - registry of routine practice.

SUMMARY:
The goal of this registry is to learn how the Medtronic Evolut™ FX+ transcatheter aortic valve implantation (TAVI) System performs in adults with severe, symptomatic aortic stenosis who need valve replacement.

The main questions it aims to answer are:

* Can using a standardized procedure for the impantation of the Medtronic Evolut™ FX+ TAVI System increase safety and efficiency?
* What are the short-term (30 days) and long-term (1 year) patient outcomes, including the need for a pacemaker, complications, and valve function?

Participants will undergo TAVI with the Medtronic Evolut™ FX+ TAVI System as part of their routine care.

Be followed during their hospital stay, at 30 days, and at 1 year to check heart health, valve function, and recovery. 500 people at 12 hospitals in Portugal will take part in this registry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects more than 18 years old, able to provide an Informed Consent:
* Severe symptomatic (defined as New York Heart Association (NYHA) class ≥ II) aortic stenosis (AS), including but not limited to: Dyspnea at rest or on exertion, fatigue, angina, syncope in the absence of another identifiable cause;
* Subjects provided written Informed Consent as approved by the Ethics Committee (EC);

Exclusion Criteria:

* Subjects with pre-existing surgical bioprosthetic aortic valve;
* Hepatic insufficiency (Child-Pugh Class B or C);
* Contraindicated for treatment with the Medtronic Evolut™ FX+ TAVU System in accordance with the Instructions for Use (IFU);
* Anatomically considered not suitable for the Medtronic Evolut™ FX+ TAVI system;
* Subjects are currently participating in another clinical investigation that may confound the results of this Registry;
* Subjects have an expected survival less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with severe, symptomatic AS with indication for TAVI, who meet the criteria for use of the Medtronic EvolutTM FX+ System in accordance with IFU and local regulations.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
VARC-3 technical success | Immediately after the index procedure
  A composite outcome assessed immediately after the TAVI procedure, including: survival, successful vascular access and device deployment/retrieval, correct positioning of a single valve, and freedom from major complications or need for surgery/intervention (excluding pacemaker).

SECONDARY OUTCOMES:
Rate of Permanent Pacemaker Implantation (PPI) | 30 days after procedure
  Percentage of participants who require a new permanent pacemaker due to new or worsening conduction disturbances.
Length of Hospital Stay | Up to 30 days after procedure
  Number of days from TAVI procedure to discharge.
All-Cause Mortality | 30 days and 1 year
  Death from any cause.
Stroke | 30 days and 1 year
  Any new neurologic deficit classified as a stroke by clinical evaluation.
Life-Threatening Bleeding | 30 days and 1 year
  Severe bleeding events defined by VARC-3 criteria.
Acute Kidney Injury | 30 days and 1 year
  Kidney dysfunction as defined by VARC-3 criteria.
Coronary Artery Obstruction | 30 days and 1 year
  Blockage requiring clinical intervention.
Major Vascular Complications | 30 days and 1 year
  Serious vascular complications as defined by VARC-3 criteria
Valve Dysfunction Requiring Reintervention | 30 days and 1 year
  Prosthetic valve dysfunction that requires repeat procedure.
Rehospitalization | 30 days and 1 year
  Rehospitalization for valve-related symptoms or worsening heart failure.
Prosthetic Valve Function | 30 days and 1 year
  Echocardiographic measures of valve function: left ventricular ejection fraction, peak velocity, mean gradient, effective orifice area, indexed effective orifice area, and prosthetic aortic valve regurgitation.
  It is defined as YES if: peak velocity is < 3 m/s AND mean gradient < 20 mmHg AND DVI > 0,25* AND Regurgitation < moderate (this means that LV and index EOA are indirectly in it, no cutt offs are needed)
  * DVI is the ratio of the Velocity-Time Integral (VTI) in the Left Ventricular Outflow Tract (LVOT) to the VTI across the stenotic aortic valve. It is measured based on the peak velocity /Grad, Effective orifice area (cm²)

OTHER OUTCOMES:
Procedural Technique Compliance (TAVI.PTrainer Survey) | During the index procedure
  Assessment of operator adherence to standardized TAVI procedural steps, including Cusp Overlap Technique, using a dedicated checklist tool.
Correlation of Procedural Compliance with Clinical Outcomes | Procedure through 1 year
  Analysis of whether higher compliance with optimized TAVI procedural steps is associated with better patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rui C Teles, MD, PhD, Principal Investigator — Hospital de Santa Cruz - Unidade Local de Saúde de Lisboa Ocidental
Locations (12):
- Portugal (12):
  - Hospitais da Universidade de Coimbra, Coimbra, Coimbra District
  - Hospital da Luz Coimbra, Coimbra, Coimbra District
  - Hospital CUF Tejo, Lisbon, Lisbon District
  - Hospital de Santa Cruz, Lisbon, Lisbon District
  - Hospital Lusíadas Lisboa, Lisbon, Lisbon District
  - Hospital da Luz Lisboa, Lisbon, Lisbon District
  - Hospital Santa Maria, Lisbon, Lisbon District
  - Hospital Santa Marta, Lisbon, Lisbon District
  - Hospital Dr. Nélio Mendonça, Funchal, Madeira
  - Hospital Universitário de São João, Porto, Porto District
  - Hospital Eduardo Santos Silva, Vila Nova de Gaia, Vila Nova de Gaia
  - Hospital do Espírito Santo de Évora, Evora, Évora District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Background] Popma JJ, Reardon MJ. Transcatheter Aortic-Valve Replacement in Low-Risk Patients. Reply. N Engl J Med. 2019 Aug 15;381(7):685. doi: 10.1056/NEJMc1908500. No abstract available. PMID 31412190
- [Background] Guerreiro C, Ferreira PC, Teles RC, Braga P, Canas da Silva P, Patricio L, Silva JC, Baptista J, de Sousa Almeida M, Gama Ribeiro V, Silva B, Brito J, Infante Oliveira E, Cacela D, Madeira S, Silveira J. Short and long-term clinical impact of transcatheter aortic valve implantation in Portugal according to different access routes: Data from the Portuguese National Registry of TAVI. Rev Port Cardiol (Engl Ed). 2020 Dec;39(12):705-717. doi: 10.1016/j.repc.2020.02.014. Epub 2020 Nov 28. English, Portuguese. PMID 33261991
- [Background] Urena M, Hayek S, Cheema AN, Serra V, Amat-Santos IJ, Nombela-Franco L, Ribeiro HB, Allende R, Paradis JM, Dumont E, Thourani VH, Babaliaros V, Francisco Pascual J, Cortes C, Del Blanco BG, Philippon F, Lerakis S, Rodes-Cabau J. Arrhythmia burden in elderly patients with severe aortic stenosis as determined by continuous electrocardiographic recording: toward a better understanding of arrhythmic events after transcatheter aortic valve replacement. Circulation. 2015 Feb 3;131(5):469-77. doi: 10.1161/CIRCULATIONAHA.114.011929. Epub 2014 Dec 2. PMID 25466975
- [Background] Auffret V, Puri R, Urena M, Chamandi C, Rodriguez-Gabella T, Philippon F, Rodes-Cabau J. Conduction Disturbances After Transcatheter Aortic Valve Replacement: Current Status and Future Perspectives. Circulation. 2017 Sep 12;136(11):1049-1069. doi: 10.1161/CIRCULATIONAHA.117.028352. PMID 28893961
- [Background] Pagnesi M, Kim WK, Baggio S, Scotti A, Barbanti M, De Marco F, Adamo M, Eitan A, Estevez-Loureiro R, Conradi L, Toggweiler S, Mylotte D, Veulemans V, Sondergaard L, Wolf A, Giannini F, Maffeo D, Pilgrim T, Montorfano M, Zweiker D, Ferlini M, Kornowski R, Hildick-Smith D, Taramasso M, Abizaid A, Schofer J, Sinning JM, Van Mieghem NM, Wohrle J, Khogali S, Van der Heyden JAS, Wood DA, Ielasi A, MacCarthy P, Brugaletta S, Hamm CW, Costa G, Testa L, Massussi M, Alarcon R, Schafer U, Brunner S, Reimers B, Lunardi M, Zeus T, Vanhaverbeke M, Naber CK, Di Ienno L, Buono A, Windecker S, Schmidt A, Lanzillo G, Vaknin-Assa H, Arunothayaraj S, Saccocci M, Siqueira D, Brinkmann C, Sedaghat A, Ziviello F, Seeger J, Rottbauer W, Brouwer J, Buysschaert I, Jelisejevas J, Bharucha A, Regueiro A, Metra M, Colombo A, Latib A, Mangieri A. Incidence, Predictors, and Prognostic Impact of New Permanent Pacemaker Implantation After TAVR With Self-Expanding Valves. JACC Cardiovasc Interv. 2023 Aug 28;16(16):2004-2017. doi: 10.1016/j.jcin.2023.05.020. Epub 2023 Jul 19. PMID 37480891
- [Background] Szotek M, Druzbicki L, Sabatowski K, Amoroso GR, De Schouwer K, Matusik PT. Transcatheter Aortic Valve Implantation and Cardiac Conduction Abnormalities: Prevalence, Risk Factors and Management. J Clin Med. 2023 Sep 19;12(18):6056. doi: 10.3390/jcm12186056. PMID 37762995
- [Background] Jorgensen TH, De Backer O, Gerds TA, Bieliauskas G, Svendsen JH, Sondergaard L. Mortality and Heart Failure Hospitalization in Patients With Conduction Abnormalities After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2019 Jan 14;12(1):52-61. doi: 10.1016/j.jcin.2018.10.053. PMID 30621978
- [Background] Maier O, Piayda K, Afzal S, Polzin A, Westenfeld R, Jung C, Zeus T, Antoch G, Kelm M, Veulemans V. Computed tomography derived predictors of permanent pacemaker implantation after transcatheter aortic valve replacement: A meta-analysis. Catheter Cardiovasc Interv. 2021 Nov 15;98(6):E897-E907. doi: 10.1002/ccd.29805. Epub 2021 Jun 2. PMID 34076343
- [Background] Abdelshafy M, Elkoumy A, Elzomor H, Abdelghani M, Campbell R, Kennedy C, Kenny Gibson W, Fezzi S, Nolan P, Wagener M, Arsang-Jang S, Mohamed SK, Mostafa M, Shawky I, MacNeill B, McInerney A, Mylotte D, Soliman O. Predictors of Conduction Disturbances Requiring New Permanent Pacemaker Implantation following Transcatheter Aortic Valve Implantation Using the Evolut Series. J Clin Med. 2023 Jul 22;12(14):4835. doi: 10.3390/jcm12144835. PMID 37510950
- [Background] Jung S, Kondruweit M, Marwan M, Achenbach S. Anatomical and Functional Predictors of Permanent Pacemaker Implantation After Transcatheter Aortic Valve Implantation. J Am Heart Assoc. 2025 May 20;14(10):e039020. doi: 10.1161/JAHA.124.039020. Epub 2025 May 15. PMID 40371597
- [Background] Jang SJ, Chen YH, Shen TC. Pitfalls in recapture or repositioning of Evolut system using cusp overlap technique. Eur Heart J. 2022 May 1;43(17):1684. doi: 10.1093/eurheartj/ehab824. No abstract available. PMID 34864965
- [Background] Wienemann H, Maier O, Beyer M, Portratz M, Tanaka T, Mauri V, Ernst A, Waldschmidt L, Kuhn E, Bleiziffer S, Wilde N, Schaefer A, Zeus T, Baldus S, Zimmer S, Veulemans V, Rudolph TK, Adam M. Cusp overlap versus standard three-cusp technique for self-expanding Evolut transcatheter aortic valves. EuroIntervention. 2023 Jun 5;19(2):e176-e187. doi: 10.4244/EIJ-D-22-01030. PMID 37013922
- [Background] Moura AR, Rodrigues JA, Braga P, Melica B, Santos L, Pires-Morais G, Sampaio F, Fontes-Carvalho R. Impact of the use of cusp-overlap projection on the incidence of permanent pacemaker implantation post-transcatheter aortic valve implantation with self-expanding valves. Rev Port Cardiol. 2023 Sep;42(9):759-769. doi: 10.1016/j.repc.2022.10.011. Epub 2023 Mar 21. English, Portuguese. PMID 36948457
- [Background] Ochiai T, Yamanaka F, Shishido K, Moriyama N, Komatsu I, Yokoyama H, Miyashita H, Sato D, Sugiyama Y, Hayashi T, Yamashita T, Tobita K, Matsumoto T, Mizuno S, Tanaka Y, Murakami M, Takahashi S, Makkar R, Saito S. Impact of High Implantation of Transcatheter Aortic Valve on Subsequent Conduction Disturbances and Coronary Access. JACC Cardiovasc Interv. 2023 May 22;16(10):1192-1204. doi: 10.1016/j.jcin.2023.03.021. PMID 37225290
- [Background] Sa MP, Van den Eynde J, Jacquemyn X, Erten O, Dokollari A, Sicouri S, Ramlawi B. Cusp-overlap versus coplanar view in transcatheter aortic valve implantation with self-expandable valves: A meta-analysis of comparative studies. Catheter Cardiovasc Interv. 2023 Feb;101(3):639-650. doi: 10.1002/ccd.30562. Epub 2023 Jan 19. PMID 36655511
- [Background] Sugiyama Y, Miyashita H, Yokoyama H, Ochiai T, Shishido K, Jalanko M, Yamanaka F, Vahasilta T, Saito S, Laine M, Moriyama N. Risk Assessment of Permanent Pacemaker Implantation After Transcatheter Aortic Valve Implantation in Patients With Preexisting Right Bundle Branch Block. Am J Cardiol. 2024 Feb 15;213:151-160. doi: 10.1016/j.amjcard.2023.12.004. Epub 2023 Dec 15. PMID 38103766
- [Background] Hazique M, Jafar Z, Lohana S, Reyaz I, Burhan M, Narayan R, Alraies MC. The Cusp Overlap Technique Reduces Pacemaker Implantation in TAVR: A Systematic Review and Meta-analysis. Am J Cardiol. 2025 Nov 1;254:75-84. doi: 10.1016/j.amjcard.2025.06.024. Epub 2025 Jun 27. PMID 40582541
- [Background] Maeno Y, Abramowitz Y, Kawamori H, Kazuno Y, Kubo S, Takahashi N, Mangat G, Okuyama K, Kashif M, Chakravarty T, Nakamura M, Cheng W, Friedman J, Berman D, Makkar RR, Jilaihawi H. A Highly Predictive Risk Model for Pacemaker Implantation After TAVR. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt A):1139-1147. doi: 10.1016/j.jcmg.2016.11.020. Epub 2017 Apr 12. PMID 28412434
- [Background] Ben-Shoshan J, Alosaimi H, Lauzier PT, Pighi M, Talmor-Barkan Y, Overtchouk P, Martucci G, Spaziano M, Finkelstein A, Gada H, Piazza N. Double S-Curve Versus Cusp-Overlap Technique: Defining the Optimal Fluoroscopic Projection for TAVR With a Self-Expanding Device. JACC Cardiovasc Interv. 2021 Jan 25;14(2):185-194. doi: 10.1016/j.jcin.2020.10.033. PMID 33478635
- [Background] Simonato M, Webb J, Kornowski R, Vahanian A, Frerker C, Nissen H, Bleiziffer S, Duncan A, Rodes-Cabau J, Attizzani GF, Horlick E, Latib A, Bekeredjian R, Barbanti M, Lefevre T, Cerillo A, Hernandez JM, Bruschi G, Spargias K, Iadanza A, Brecker S, Palma JH, Finkelstein A, Abdel-Wahab M, Lemos P, Petronio AS, Champagnac D, Sinning JM, Salizzoni S, Napodano M, Fiorina C, Marzocchi A, Leon M, Dvir D. Transcatheter Replacement of Failed Bioprosthetic Valves: Large Multicenter Assessment of the Effect of Implantation Depth on Hemodynamics After Aortic Valve-in-Valve. Circ Cardiovasc Interv. 2016 Jun;9(6):e003651. doi: 10.1161/CIRCINTERVENTIONS.115.003651. PMID 27301396
- [Background] Testa L, Latib A, Brambilla N, De Marco F, Fiorina C, Adamo M, Giannini C, Angelillis M, Barbanti M, Sgroi C, Poli A, Ferrara E, Bruschi G, Russo CF, Matteo M, De Felice F, Musto C, Curello S, Colombo A, Tamburino C, Petronio AS, Bedogni F. Long-term clinical outcome and performance of transcatheter aortic valve replacement with a self-expandable bioprosthesis. Eur Heart J. 2020 May 21;41(20):1876-1886. doi: 10.1093/eurheartj/ehz925. PMID 31904800
- [Background] Trimaille A, Carmona A, Hmadeh S, Truong DP, Marchandot B, Kikuchi S, Matsushita K, Ohlmann P, Schini-Kerth V, Rodes-Cabau J, Pibarot P, Morel O. Transcatheter Aortic Valve Durability: Focus on Structural Valve Deterioration. J Am Heart Assoc. 2025 Jul;14(13):e041505. doi: 10.1161/JAHA.125.041505. Epub 2025 Jun 18. PMID 40530490
- [Background] Van Belle E, Teles RC, Pyxaras SA, Kalpak O, Johnson TW, Barbash IM, De Luca G, Kostov J, Parma R, Vincent F, Brugaletta S, Debry N, Toth GG, Ghazzal Z, Deharo P, Milasinovic D, Kaspar K, Saia F, Mauri Ferre J, Kammler J, Muir DF, O'Connor S, Mehilli J, Thiele H, Weilenmann D, Witt N, Joshi F, Kharbanda RK, Piroth Z, Wojakowski W, Geppert A, Di Gioia G, Pires-Morais G, Petronio AS, Estevez-Loureiro R, Ruzsa Z, Kefer J, Kunadian V, Van Mieghem N, Windecker S, Baumbach A, Haude M, Dudek D. EAPCI Core Curriculum for Percutaneous Cardiovascular Interventions (2020): Committee for Education and Training European Association of Percutaneous Cardiovascular Interventions (EAPCI). A branch of the European Society of Cardiology. EuroIntervention. 2021 May 17;17(1):23-31. doi: 10.4244/EIJ-D-18-00448. PMID 32624457
- [Background] Teles RC, Van Belle E, Parma R, Tarantini G, van Mieghem N, Mylotte D, Silva JD, O'Connor S, Sondegaard L, Luz A, Amat-Santos IJ, Arzamendi D, Blackman D, De Backer O, Kunadian V, Buchanan GL, MacCarthy P, Lurz P, Naber C, Chieffo A, Paradies V, Gilard M, Vincent F, Fraccaro C, Mehilli J, Giannini C, Silva B, Poliacikova P, Karam N, Veulemans V, Thiele H, Pilgrim T, van Wely M, James S, Schmidt MR, Uebing A, Ruck A, Ghanem A, Ghazzal Z, Joshi FR, Favero L, Hermanides R, Ninios V, Fovino LN, Nuis RJ, Deharo P, Kala P, Elbaz-Greener G, Tchetche D, Agricola E, Thielmann M, Donal E, Bonaros N, Droogmans S, Czerny M, Baumbach A, Barbato E, Dudek D. Percutaneous Valvular and Structural Heart Disease Interventions. 2024 Core Curriculum of the European Association of Percutaneous Cardiovascular Interventions (EAPCI) of the ESC in collaboration with the European Association of Cardiovascular Imaging (EACVI) and the Cardiovascular Surgery Working Group (WG CVS) of the European Society of Cardiology. EuroIntervention. 2024 Aug 30;20(22):1370-9. doi: 10.4244/EIJ-D-23-00983. Online ahead of print. PMID 39207816
- [Background] Grubb KJ, Gada H, Mittal S, Nazif T, Rodes-Cabau J, Fraser DGW, Lin L, Rovin JD, Khalil R, Sultan I, Gardner B, Lorenz D, Chetcuti SJ, Patel NC, Harvey JE, Mahoney P, Schwartz B, Jafar Z, Wang J, Potluri S, Vora AN, Sanchez C, Corrigan A, Li S, Yakubov SJ. Clinical Impact of Standardized TAVR Technique and Care Pathway: Insights From the Optimize PRO Study. JACC Cardiovasc Interv. 2023 Mar 13;16(5):558-570. doi: 10.1016/j.jcin.2023.01.016. PMID 36922042
- [Background] Grubb KJ, Gada H, Fraser D, Rodes-Cabau J, Nazif TM, Mittal S, Dvir D, Teiger E, Lin L, Rovin JD, Khalil RF, Sultan I, Yudi MB, Gardner B, Lorenz D, Chetcuti S, Patel NC, Harvey J, Mahoney P, Talreja D, Trani C, Mylotte D, Schwartz B, Jafar Z, Van der Heyden J, Maffeo D, Yong G, Moris C, Wang J, Gooley R, Flor K, Yeh YJ, Yakubov SJ. Global Results From the Optimize PRO Study: Standardized TAVR Technique and Care Pathway. J Soc Cardiovasc Angiogr Interv. 2025 May 1;4(5):103515. doi: 10.1016/j.jscai.2025.103515. eCollection 2025 May. PMID 40454273
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579
- [Background] Wassef AWA, Rodes-Cabau J, Liu Y, Webb JG, Barbanti M, Munoz-Garcia AJ, Tamburino C, Dager AE, Serra V, Amat-Santos IJ, Alonso Briales JH, San Roman A, Urena M, Himbert D, Nombela-Franco L, Abizaid A, de Brito FS Jr, Ribeiro HB, Ruel M, Lima VC, Nietlispach F, Cheema AN. The Learning Curve and Annual Procedure Volume Standards for Optimum Outcomes of Transcatheter Aortic Valve Replacement: Findings From an International Registry. JACC Cardiovasc Interv. 2018 Sep 10;11(17):1669-1679. doi: 10.1016/j.jcin.2018.06.044. PMID 30190058